CLINICAL TRIAL: NCT04006327
Title: Demoralization Among Palliative Care Patients and Their Family Caregivers in Hong Kong: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hospital Authority of Hong Kong (Bradbury Hospice) (Unknown)
Responsible Party: Principal Investigator, Wallace Chi Ho Chan, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2018.448
Record Dates: First submitted 2019-03-25; First posted 2019-07-05 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Demoralization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative care patients and their family caregivers: The present study is a cross-sectional study with single group study design. Only palliative care patients and their family caregivers will be recruited.
  Interventions: Other: No intervention will be provided as this study is a cross-sectional observational study.

INTERVENTIONS:
Other: No intervention will be provided as this study is a cross-sectional observational study. — This item is not applicable because this study is a cross-sectional observational study and no intervention will be provided to participants.

SUMMARY:
This study aims to explore the prevalence of demoralization among palliative care patients and family caregivers in Hong Kong and examines psychosocial factors associated with demoralization. We hypothesized that higher depression, caregiving strain and caregiver support needs would lead to higher demoralization, and greater perceived family support was associated with lower demoralization among patients and family caregivers.

DETAILED DESCRIPTION:
Literature Review:

Demoralization in palliative care Palliative care patients (PCP) and their family caregivers are always confronted with death and dying issues. The nature of terminal illness may lead to their experience of demoralization. The importance of addressing the demoralization syndrome among PCP was first proposed by Clarke and Kissane (2002). A systematic review reported that the prevalence of demoralization is about 13% to 18% among palliative care patients (Robinson, Kissane, Brooker & Burney, 2016). Only one study examined the prevalence of demoralization among family caregivers of PCP and that aro10% of them suffered from moderate to severe demoralization (Hudson, Thomas, Trauer, Remedios, & Clarke, 2011).

PCP and family caregivers may find it difficult to cope with the challenges associated with the terminal illness, and that they may experience a form of existential distress, which is characterized by a sense of meaninglessness, hopelessness and helplessness (Figueriredo, 2013; Robinson, et al., 2016). Demoralization was considered as a key cause of developing suicidal ideations (Julião, Nunes & Barbosa, 2016).

Conceptualization and definition of demoralization Kissane (2000) conceptualized demoralization as a syndrome with the following diagnostic criteria: 1. The experience of emotional distress such as hopelessness and having meaning and purpose in life lost; 2. Attitudes of helplessness, failure, pessimism, and lack of a worthwhile future; 3. Reduced coping to respond differently; 4. Social isolation and deficiencies in social support; 5.Persistence if the above-mentioned phenomena across 2 or more weeks; and 6. Features of major depression have not superseded as the primary disorder (Robinson et al., 2016, p.96). Demoralization should be differentiated from depression, e.g. demoralized patients may still enjoy the present moment but feel despair towards future (Clarke & Kissane, 2002; Kissane & Doolittle, 2015). Demoralization may exist independently but can also co-exist with depression. Previous studies showed that 14-27.4% of patients were demoralized but not depressive, while 21.7-33% patients experienced both demoralization and depression (Fang et al., 2014).

Factors associated with demoralization Previous studies showed that demoralization was associated with various socio-economic, physical and psychosocial factors. High demoralization was associated with reduced quality of life, emotional and existential distress (e.g. depression, anxiety and desire for hastened death, hopelessness, helplessness and loss of meaning) and declining physiological functions (e.g. pain, fatigue and sleep disorders) (Robinson, Kissane, Brooker & Burney, 2015; Tang, Wang & Chou, 2015). A strong relationship was also found between demoralization and social functioning (Kissane and Doolittle, 2015; Robinson et al., 2015; Tang et. al, 2015). Furthermore, demoralization was found associated with sociodemographic, spiritual and familial factors, such as unemployment, sex, family dysfunction, spiritual problem and dimensions to a person's life (Lee et al., 2011; Li et al, 2017; Kissane and Doolittle, 2015; Robinson et al., 2015).

Demoralization has been studied in the western societies in the past decade but little has been known about demoralization prevalence among palliative care patients and family caregivers in Hong Kong. As demoralization is a newly introduced concept, there is limited understanding on its epidemiology and how it can be minimized among PC patients and caregivers. It is thus important to conduct a pilot study in Hong Kong to explore the prevalence of demoralization and factors associated with demoralization.

Objectives:

1. To explore the prevalence of demoralization among palliative care patients and their family caregiver in Hong Kong;
2. To examine the relationships of demoralization with different psychosocial factors (e.g. depression, perceived family support, caregiving strain) among palliative care patients and family caregivers in Hong Kong;
3. To understand how the illness experience may lead to demoralization among palliative care patients and their family caregivers in Hong Kong;
4. To understand how palliative care may reduce demoralization among palliative care patients and their family caregivers in Hong Kong;
5. To understand how palliative care patients and family caregivers care may cope with the illness to avoid demoralization

Methods:

This study targets to recruit 200 palliative care patients (PCP) and family caregivers who are newly referred to the Medical Social work department of Bradbury Hospice. This study will employ a mixed method design to achieve the study objectives.

For quantitative arm, patients and caregivers will be asked to complete a survey respectively, which include different validated instruments. Assistance will be given for completing the survey if necessary. For patient questionnaire, we will include the Chinese version of Demoralization Scale (Hung et al., 2010), the 10-item version of Center for Epidemiological Studies Depression (CES-D), and the Family subscale of the Chinese version of Multidimensional Scale of Perceived Social Support. For the caregiver's questionnaire, similar to the patient questionnaire, we plan to include the Demoralization Scale and CES-D, but we also include the Chinese version of Modified Caregivers' Strain Index and the Carer Support Needs Assessment tool (CSNAT). A total of 200 patients and caregivers will be recruited. Data will be entered into SPSS for analysis.

For qualitative arm, individual interviews will be conducted with PCP and caregivers by a trained research assistant. 6 PCP and 6 family caregivers will be purposively selected for interview based on their demoralization level which was reflected from their demoralization scores in the quantitative data. (i.e. 3 patients and 3 family caregivers from each of the following groups: Low demoralization and high demoralization group).

Data Management and analysis:

All data will be stored confidentially in order to protect participant's privacy. Quantitative data will be entered to SPSS for data analysis. Descriptive, bivariate correlations bivariate correlations and regression analysis will be conducted and missing data will be handled by mean substitution. For interviews data, all the audio-recorded interviews will be transcribed to text for data analysis. Thematic analysis will be conducted to identify the key themes.

ELIGIBILITY:
For palliative care patients

Inclusion Criteria:

* Must be currently living in the community
* Chinese who are able to communicate in Cantonese

Exclusion Criteria:

-Patients who are assessed by social workers as emotionally too distressful for participating in the research.

For caregivers

Inclusion criteria:

-Caregivers must be the primary family caregivers of the patients

Exclusion criteria:

-Caregivers who are assessed by social workers as emotionally too distressful for participating in the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study targets palliative care patients of Bradbury Hospice (BBH) and their family caregivers who are newly referred to the Medical Social Work Department of Bradbury Hospice.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Demoralization of patients and caregivers | This is a one-time self-reported assessment which will take less than 15 minutes to complete.
  Demoralization of patients and caregivers will be measured by the Chinese version of Demoralization Scale (DS).The instrument comprises of 24 items and each item is rated on a 4-point Likert-type scale that ranged from 1 (very disagreed) to 5 (very agreed). Items for each responses will be summed up to create a total score ranging from 0 to 30. The DS also provides 5 subscores, namely, loss of meaning and purpose, dysphoria, disheartenment, helplessness and sense of failure. A higher total score indicates a higher level of demoralization

SECONDARY OUTCOMES:
Depression of patients and caregivers | This is a one-time self-reported assessment which will take less than 15 minutes to complete.
  The depressive symptoms of patients and caregivers will be measured by the ten-item Chinese version of Center for Epidemiological Studies Depression scale (CESD-10), which is a self-reported measurement on depression containing 10 items. Ratings were based on a 4-point Likert scale ranging from 0 (rarely or none of the time) to 3 (most or all of the time). Items for each responses will be summed up to create a total score ranging from 0 to 30. A higher CESD score indicates a higher level of depression.
Perceived Family Support of patients | This is a one-time self-reported assessment which will take less than 15 minutes to complete.
  Perceived family support of patients will be measured by the family subscale of the Chinese version of Multidimensional scale of perceived social support. This scale contains 13 items and rating was based on a 4 point Likert scale ranging from 1 (very disagreed) to 4 (Very agreed). Items for each responses will be summed up to create a total score of family support ranging from 13 to 52. A higher family subscale score indicates a higher level of perceived support from family.
Caregiver Strain of caregivers | This is a one-time self-reported assessment which will take less than 15 minutes to complete.
  Caregiver strain of caregivers will be measured with the Chinese version of Modified caregiver strain index (M-CSI). The scale comprises of 13 items that measure strain related to care provision. Caregivers will be asked to indicate the level of distress caused by each item, ranging from "not at all" to "Yes, quite often," on a scale of 0 to 2. A total strain score will be obtained by adding up the scores for each response, with a possible total score ranging from 0 to 26. A higher score indicates higher level of caregiver strain.
Caregiver Support Needs of caregivers | This is a one-time self-reported assessment which will take less than 15 minutes to complete.
  Caregiver Support needs of family caregivers will be measured by the Chinese version of caregivers support needs assessment tool (CSNAT). The CSNAT was originally designed as a screening tool to identify caregivers key support needs that require further supports. This tool contains 14 support domains and there are 4 response options for each of the CSNAT items, which allows family caregivers to indicate the extent of their support requirements for each domain: "no more", "a little more," "quite a bit more," or "very much more". This assessment tool does not create a total score of caregiver support needs.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Ho Wallace Chan, BSoc, Ph.D, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Bradbury Hospice (BBH), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke DM, Kissane DW. Demoralization: its phenomenology and importance. Aust N Z J Psychiatry. 2002 Dec;36(6):733-42. doi: 10.1046/j.1440-1614.2002.01086.x. PMID 12406115
- [Background] Fang CK, Chang MC, Chen PJ, Lin CC, Chen GS, Lin J, Hsieh RK, Chang YF, Chen HW, Wu CL, Lin KC, Chiu YJ, Li YC. A correlational study of suicidal ideation with psychological distress, depression, and demoralization in patients with cancer. Support Care Cancer. 2014 Dec;22(12):3165-74. doi: 10.1007/s00520-014-2290-4. Epub 2014 Jun 17. PMID 24935648
- [Background] Figueiredo JMD. Distress, demoralization and psychopathology: diagnostic boundaries. Eur J Psychiatry. 2013; 27(1): 61-73.
- [Background] Hudson PL, Thomas K, Trauer T, Remedios C, Clarke D. Psychological and social profile of family caregivers on commencement of palliative care. J Pain Symptom Manage. 2011 Mar;41(3):522-34. doi: 10.1016/j.jpainsymman.2010.05.006. Epub 2010 Dec 3. PMID 21123026
- [Background] Hung HC, Chen HW, Chang YF, Yang YC, Liu CL, Hsieh RK, ... & Liu SI. Evaluation of the reliability and validity of the Mandarin Version of Demoralization Scale for cancer patients. J Intern Med Taiwan. 2010; 21(6): 427-435.
- [Background] Juliao M, Nunes B, Barbosa A. Prevalence and factors associated with demoralization syndrome in patients with advanced disease: Results from a cross-sectional Portuguese study. Palliat Support Care. 2016 Oct;14(5):468-73. doi: 10.1017/S1478951515001364. Epub 2016 Jan 6. PMID 26732616
- [Background] Kissane DW. Psychospiritual and existential distress. The challenge for palliative care. Aust Fam Physician. 2000 Nov;29(11):1022-5. PMID 11127057
- [Background] Lee CY, Fang CK, Yang YC, Liu CL, Leu YS, Wang TE, Chang YF, Hsieh RK, Chen YJ, Tsai LY, Liu SI, Chen HW. Demoralization syndrome among cancer outpatients in Taiwan. Support Care Cancer. 2012 Oct;20(10):2259-67. doi: 10.1007/s00520-011-1332-4. Epub 2011 Nov 27. PMID 22120003
- [Background] Li YC, Ho CH, Wang HH. Protective Factors of Demoralization among Cancer Patients in Taiwan: An Age-matched and Gender-matched Study. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Sep;11(3):174-179. doi: 10.1016/j.anr.2017.07.001. Epub 2017 Aug 10. PMID 28991597
- [Background] Robinson S, Kissane DW, Brooker J, Burney S. A systematic review of the demoralization syndrome in individuals with progressive disease and cancer: a decade of research. J Pain Symptom Manage. 2015 Mar;49(3):595-610. doi: 10.1016/j.jpainsymman.2014.07.008. Epub 2014 Aug 15. PMID 25131888
- [Background] Robinson S, Kissane DW, Brooker J, Burney S. A Review of the Construct of Demoralization: History, Definitions, and Future Directions for Palliative Care. Am J Hosp Palliat Care. 2016 Feb;33(1):93-101. doi: 10.1177/1049909114553461. Epub 2014 Oct 7. PMID 25294224
- [Background] Tang PL, Wang HH, Chou FH. A Systematic Review and Meta-Analysis of Demoralization and Depression in Patients With Cancer. Psychosomatics. 2015 Nov-Dec;56(6):634-43. doi: 10.1016/j.psym.2015.06.005. Epub 2015 Jun 19. PMID 26411374